CLINICAL TRIAL: NCT03814486
Title: Etude Descriptive Retrospective de la Transfusion Plaquettaire Chez Des Patients Atteints d'hémopathie Maligne en Phase Palliative et Suivis au CHU de Besançon
Brief Title: Retrospective Descriptive Study of Platelet Transfusion in Patients With Palliative Hematologic Malignancies at the University Hospital of Besançon
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: J Moracchini
Record Dates: First submitted 2019-01-02; First posted 2019-01-24 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-12

CONDITIONS: Platelet Transfusion; Palliative Care
Keywords: platelet transfusion; palliative care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient transfused in platelet in the 6 last months of life: patient with hematological malignancies follow or hospitalised at least once in CHU of Besancon died in the period of the study transfused at least once in the 6 months of life
  Interventions: Other: descriptive

INTERVENTIONS:
Other: descriptive — evaluate in number and efficacy platelet transfusion at the end of life, demographic characteristic are also noted

SUMMARY:
Development of palliative care is less effective for patients with hematologic malignancies. Limited data is available for end of life care in this population, moreover with thrombocytopenic patients. Thrombopenia is a frequent complication, specific of bone marrow involvement in those diseases or its treatments. Yet, a few studies was interested in, whereas platelet transfusion is the only treatment indicated. As it represent a scarce, limited resource, the ethical principles are in conflict in this setting.

The purpose of this study was to describe retrospectively platelet transfusion in the six last few month of life of patients with hematologic malignancies at the CHU of Besançon (France) between 01/07/15 and 31/12/16.

ELIGIBILITY:
Inclusion Criteria:

* patient with hematological malignancies
* transfused in platelet at least once in the last 6 months of life
* hospitalised or follow up at the CHU of Besancon at least once
* dead during the period of the study

Exclusion Criteria:

* patient with other oncologic malignancies
* not transfused in platelet in the last 6 months of life
* never hospitalised or follow up at the CHU of Besancon
* alive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with hematological malignancies,transfused in platelet at least once in the last 6 months of life, hospitalised or follow up at the CHU of Besancon at least once and dead during the period of the study
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
evaluate frequency of platelet transfusion at the end of life | 18 months (between 07/01/2015 and 12/31/2016)
  to calculate the number of platelet transfusion at the end of life. The number of platelet transfusion between 6 months and death are collected in each periods of 2 weeks to calculate the number of transfusion per patient during each 2 weeks.
evaluate efficacy of prophylactic platelet transfusion at the end of life | 18 months (between 07/01/2015 and 12/31/2016)
  to calculate the platelet yield in percentage
evaluate efficacy of non prophylactic platelet transfusion at the end of life | 18 month (between 07/01/2015 and 12/31/2016)
  to calculate the transfusional interval between 2 platelet transfusion in days

SECONDARY OUTCOMES:
demographic characteristic | 18 months (between 07/01/2015 and 12/31/2016)
  characteristic of patient (age, diagnosis,location of death, palliative care received...)

CONTACTS AND LOCATIONS:
Overall Officials: regis aubry, ph, Study Director — Centre Hospitalier Universitaire de Besancon
Locations (1):
- Moracchini, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided
patient were dead during the period of recruitment. Characteristic of patient could be used for other purpose

REFERENCES:
- [Background] Hochsmann B, Moicean A, Risitano A, Ljungman P, Schrezenmeier H. Supportive care in severe and very severe aplastic anemia. Bone Marrow Transplant. 2013 Feb;48(2):168-73. doi: 10.1038/bmt.2012.220. Epub 2012 Dec 3. PMID 23208312
- [Background] Sherbeck JP, Boss RD. Ethical Questions about Platelet Transfusions at the End of Life. AMA J Ethics. 2016 Aug 1;18(8):764-70. doi: 10.1001/journalofethics.2016.18.8.ecas1-1608. PMID 27550559
- [Background] Salacz ME, Lankiewicz MW, Weissman DE. Management of thrombocytopenia in bone marrow failure: a review. J Palliat Med. 2007 Feb;10(1):236-44. doi: 10.1089/jpm.2006.0126. PMID 17298272
- [Background] Lassauniere JM, Bertolino M, Hunault M, Zittoun R, Verspieren P, Moh-Klaren J, Jaulmes D, Colombat P. Platelet transfusions in advanced hematological malignancies: a position paper. J Palliat Care. 1996 Spring;12(1):38-41. PMID 8857246
- [Background] Boggs DR. Jehovah's Witnesses with leukemia. Hosp Pract (Off Ed). 1985 Mar 15;20(3):92, 94-5, 98 passim. doi: 10.1080/21548331.1985.11703015. No abstract available. PMID 2414307
- [Result] Wang WS, Ma JD, Nelson SH, Revta C, Buckholz GT, Mulroney C, Roeland EJ. Transfusion practices at end of life for hematopoietic stem cell transplant patients. Support Care Cancer. 2018 Jun;26(6):1927-1931. doi: 10.1007/s00520-017-4023-y. Epub 2017 Dec 28. PMID 29285557